CLINICAL TRIAL: NCT05744713
Title: An Observational Study of Patients With Chronic Liver Disease
Status: Enrolling by invitation | Type: Observational
Sponsor: Target PharmaSolutions, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TARGET-LD
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Liver Disease; Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole blood Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Disease Cohort
  Interventions: Other: Observational
- Engaged Cohort
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — Observational

SUMMARY:
TARGET-Liver Disease (TARGET-LD) is an observational research study to conduct a comprehensive review of outcomes for patients with chronic liver disease (CLD).

ELIGIBILITY:
Inclusion Criteria:

Disease Cohort

•Adult* patients at the time of enrollment with a diagnosis of CLD/cirrhosis by ICD-10 code in the EHR interface

Engaged Cohort

* Adult* patients diagnosed and managed for CLD/cirrhosis invited to participate
* Ability to provide written informed consent

Exclusion Criteria:

Disease Cohort

* Death
* Manual removal (sponsor or site request)
* No EHR interface encounter > 3 years.

Engaged Cohort

* Patient expressed desire to withdraw consent to complete PROs
* Failure to complete PROs within 24 weeks of initial invitation
* Greater than 24 months lapse of survey completion after baseline surveys completed
* Additionally, the criteria detailed for Disease Cohort apply to the Engaged Cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will include adults who are being managed for chronic liver disease or cirrhosis of any etiology.
Sampling Method: Non-Probability Sample
Enrollment: 500000 (Estimated)
Dates: Start 2024-02-19 (Actual); Primary Completion 2037-12-31 (Estimated); Study Completion 2037-12-31 (Estimated)

PRIMARY OUTCOMES:
To characterize the natural history of disease in patients with CLD from various etiologies and Cirrhosis | 20 Years
To assess safety and effectiveness of CLD/Cirrhosis treatments and treatments for complications of any chronic liver disease | 20 Years
To establish learning health networks focused on quality of care for patients | 20 Years

SECONDARY OUTCOMES:
To evaluate provider management practices in the treatment of patients with CLD/Cirrhosis | 20 Years
To evaluate longitudinal and patient reported outcomes in CLD/Cirrhosis | 20 Years

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Stanford Medicine, Redwood City, California
  - Georgetown Medstar Transplant Institute, Washington D.C., District of Columbia
  - Rush University Medical Center, Chicago, Illinois
  - Columbia University Irving Medical Center/ New York Presbyterian Hospital, New York, New York
  - Atrium Health Center for Liver Disease and Transplant, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Temple University - Lewis Katz School of Medicine, Philadelphia, Pennsylvania
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided